CLINICAL TRIAL: NCT02371746
Title: A Multi-Center, Three-Stage, Open-Label, Prospective, Active-Comparator-Controlled Phase 2a Study of ENV515 (Travoprost) Intracameral Implant in Patients With Bilateral Ocular Hypertension or Early Primary Open-Angle Glaucoma
Brief Title: Safety and Efficacy of ENV515 Travoprost Extended Release (XR) in Patients With Bilateral Ocular Hypertension or Primary Open Angle Glaucoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Envisia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENV515-01
Record Dates: First submitted 2015-02-20; First posted 2015-02-26 (Estimated); Results first posted 2019-10-17 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-09

CONDITIONS: Glaucoma and Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): ENV515-1 and ENV515-3 implants in Study Eye for 28 days
  Interventions: Drug: ENV515-3 Travoprost XR; Drug: ENV515-1 Travoprost XR
- Cohort 2 (Experimental): Two ENV515-3 implants in Study Eye for 12 months with optional 6 month and 3 month extensions (total of 21 months)
  Interventions: Drug: ENV515-3 Travoprost XR
- Cohort 3 (Experimental): One or two ENV515-3-2 implants in Study Eye with optional 6 months and additional 6 month extension (total of 24 months)
  Interventions: Drug: ENV515-3-2 Travoprost XR

INTERVENTIONS:
Drug: ENV515-3 Travoprost XR
  Arms: Cohort 1; Cohort 2
Drug: ENV515-1 Travoprost XR
  Arms: Cohort 1
Drug: ENV515-3-2 Travoprost XR
  Arms: Cohort 3

SUMMARY:
This is a multiple cohort study that will evaluate the safety and efficacy of ENV515 travoprost XR in patients with open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of either ocular hypertension or open angle glaucoma in both eyes.
* Are currently treated with topical PGA for ocular hypertension in both eyes.
* Patients who in the opinion of the Investigator: have an IOP in both eyes that is considered to be adequately controlled, can be safely withdrawn from IOP medications in both eyes during the washout period, and who are not considered to be at significant risk for disease progression throughout the trial.

Exclusion Criteria:

* Eye surgery (including cataract surgery) within the past 3 months.
* History of glaucoma related surgery.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-02-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Chandler, Arizona
  - Garden Grove, California
  - Inglewood, California
  - Redding, California
  - Morrow, Georgia
  - Indianapolis, Indiana
  - Chesterfield, Missouri
  - Kansas City, Missouri
  - Cincinnati, Ohio
  - Portland, Oregon
  - Sioux Falls, South Dakota
  - Austin, Texas
  - Houston, Texas
  - San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 - Group 1: 2 ENV515-3 implants (28.2 μg travoprost) in Study Eye for 28 days
- Cohort 1 - Group 2: 3 ENV515-3 implants (42.3 μg travoprost) in Study Eye for 28 days
- Cohort 1 - Group 3: 1 ENV515-1 implant (42.5 μg travoprost) in Study Eye for 28 days
- Cohort 1 - Group 4: 2 ENV515-1 implants (85.0 μg travoprost) in Study Eye for 28 days
- Cohort 2: 2 ENV515-3 implants (28.2 μg travoprost) in Study Eye for up to 21 months
- Cohort 3 - Group 1: 1 ENV515-3-2 implant (26.1 μg travoprost) in Study Eye for up to 24 months
- Cohort 3 - Group 2: 2 ENV515-3-2 implants (52.2 μg travoprost) in Study Eye for up to 24 months
Period: Overall Study
Arm/Group | Cohort 1 - Group 1 | Cohort 1 - Group 2 | Cohort 1 - Group 3 | Cohort 1 - Group 4 | Cohort 2 | Cohort 3 - Group 1 | Cohort 3 - Group 2
Started | 7 | 10 | 2 | 2 | 5 | 6 | 9
Completed | 7 | 10 | 2 | 2 | 5 | 6 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Consent withdrawn | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Cohort 1 - Group 4: 2 ENV515-3 implants (85.0 μg travoprost) in Study Eye for 28 days
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - Group 1 | Cohort 1 - Group 2 | Cohort 1 - Group 3 | Cohort 1 - Group 4 | Cohort 2 | Cohort 3 - Group 1 | Cohort 3 - Group 2 | Total
Number analyzed (Participants) | 7 | 10 | 2 | 2 | 5 | 6 | 9 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 0 | 1 | 3 | 5 | 3 | 13
  >=65 years | 7 | 9 | 2 | 1 | 2 | 1 | 6 | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Cohort 1 was analyzed separately from Cohorts 2 and 3 due to the Cohort 1 database being locked prior to the completion of Cohorts 2 and 3.
  Years
    Cohort 1: number analyzed (Participants) | 7 | 10 | 2 | 2 | 0 | 0 | 0 | 21
    Cohort 1 | 74.32 (4.729) | 71.99 (4.213) | 71.29 (7.128) | 62.46 (8.188) |  |  |  | 71.79 (5.619)
    Cohorts 2 and 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 6 | 9 | 20
    Cohorts 2 and 3 |  |  |  |  | 57.412 (11.4833) | 59.472 (7.2299) | 64.462 (10.4534) | 61.203 (9.8634)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 2 | 2 | 4 | 2 | 6 | 24
  Male | 2 | 7 | 0 | 0 | 1 | 4 | 3 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 4
  Not Hispanic or Latino | 5 | 10 | 2 | 1 | 4 | 6 | 9 | 37
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 5
  White | 7 | 7 | 2 | 2 | 5 | 5 | 7 | 35
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 10 | 2 | 2 | 5 | 6 | 9 | 41
Intraocular Pressure (mm Hg) [Mean (Standard Deviation); unit: mm Hg] — All IOPs were measured with a Goldmann applanation tonometer. Population: Cohort 1 was analyzed separately from Cohorts 2 and 3 due to the Cohort 1 database being locked prior to the completion of Cohorts 2 and 3.
  mm Hg
    Cohort 1: number analyzed (Participants) | 7 | 10 | 2 | 2 | 0 | 0 | 0 | 21
    Cohort 1 | 24.57 (2.370) | 24.12 (2.277) | 24.83 (3.064) | 26.67 (1.414) |  |  |  | 24.58 (2.267)
    Cohorts 2 and 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5 | 6 | 9 | 20
    Cohorts 2 and 3 |  |  |  |  | 26.2 (2.39) | 28.2 (2.99) | 25.2 (1.56) | 26.4 (2.50)

OUTCOME MEASURES:

1. Primary Outcome: Summary of Change From Baseline Average Intraocular Pressure Diurnal Measurement by Treatment Group Population (Cohort 1)
Description: Average intraocular pressure (IOP) diurnal measurement is calculated by taking the average of the intraocular pressure measurements at 8AM, 10AM and 4PM. The protocol was later amended (Amendment 09) to a safety only study so the diurnal measurements were no longer collected for Cohorts 2 and 3; only the 8AM IOP was collected as a safety assessment only.
Time Frame: Baseline and Day 25
Population: Safety Population
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Cohort 3 - Group 1: 1 ENV515-3-2 implant (28.2 μg travoprost) in Study Eye for for up to 24 months
Arm/Group | Cohort 1 - Group 1 | Cohort 1 - Group 2 | Cohort 1 - Group 3 | Cohort 1 - Group 4 | Cohort 2 | Cohort 3 - Group 1 | Cohort 3 - Group 2
Number analyzed (Participants) | 7 | 10 | 2 | 2 | 0 | 0 | 0
mm Hg | -5.10 (1.707) | -6.65 (2.076) | -3.17 (1.179) | -5.67 (0.000) |  |  |
Statistical Analysis 1: Comparison: Cohort 1 - Group 1 vs Cohort 1 - Group 2 vs Cohort 1 - Group 3 vs Cohort 1 - Group 4; estimatCohort 1 all Groups: Non-study eye: TRAVANTAN Z Cohort 1 - Group 1: Study Eye: 28.2 ug travoprost Cohort 1 - Group 2: Study Eye: 42.3 ug travoprost Cohort 1 - Group 3: Study Eye: 42 .5 ug travoprost Cohort 1 - Group 4: Study Eye: 85.0 ug travoprost; Test type: Superiority; p < 0.001, ANCOVA; Change from baseline = 30.4, 95% CI 2-sided [-1.8 to 36.6], Standard Deviation 1.84

ADVERSE EVENTS:
Time Frame: Cohort 1 - Adverse Events (AEs) were collected for up to 49 days post-treatment. Cohort 2 - AEs were collected for up to 12 months (+/- 7 days), 18 months (+/- 7 days) for Extension 1, and 21 months (+/- 7 days) for Extension 2 post-treatment. Cohort 3 - AEs were collected for up to 12 months (+/- 7 days), 18 months (+/- 7 days) for Extension 1, and 24 months (+/- 7 days) for Extension 2 post-treatment.
Description: In addition, the term Adverse Event of Special Interest (AESI) was used and defined to include any corneal events including corneal edema detected via slit lamp or pachymetry, corneal opacity, and any suspected changes in corneal endothelial cell counts determined by the central reading center of 30% or greater change from baseline (V2) as determined via specular microscopy. Systematic assessment included AE queries at each patient visit.
Groups:
- Cohort 2 - Group 3: 1 ENV515-1 implant (42.5 μg travoprost) in Study Eye for 28 days
Arm/Group | Cohort 1 - Group 1 | Cohort 1 - Group 2 | Cohort 2 - Group 3 | Cohort 1 - Group 4 | Cohort 2 | Cohort 3 - Group 1 | Cohort 3 - Group 2
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/10 | 0/2 | 0/2 | 0/5 | 0/6 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/7 | 1/10 | 0/2 | 0/2 | 0/5 | 0/6 | 4/9
Other Adverse Events (participants affected / at risk) | 4/7 | 7/10 | 2/2 | 2/2 | 5/5 | 6/6 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - Group 1 (N=7) | Cohort 1 - Group 2 (N=10) | Cohort 2 - Group 3 (N=2) | Cohort 1 - Group 4 (N=2) | Cohort 2 (N=5) | Cohort 3 - Group 1 (N=6) | Cohort 3 - Group 2 (N=9)
Corneal edema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Corneal endothelial cell loss (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paget's disease of the right nipple (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - Group 1 (N=7) | Cohort 1 - Group 2 (N=10) | Cohort 2 - Group 3 (N=2) | Cohort 1 - Group 4 (N=2) | Cohort 2 (N=5) | Cohort 3 - Group 1 (N=6) | Cohort 3 - Group 2 (N=9)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Meniere's disease (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anterior chamber cell (Eye disorders) | 1 | 2 | 0 | 1 | 1 | 0 | 2
Anterior chamber flare (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anterior chamber inflammation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Chalazion (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 1 | 3 | 0 | 0 | 1 | 0 | 0
Conjunctival oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Corneal edema (Eye disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0
Corneal endothelial cell loss (Eye disorders) | 0 | 1 | 0 | 0 | 2 | 2 | 4
Corneal epithelial microcysts (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Corneal opacity (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Corneal thickening (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye allergy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye inflammation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1
Eye pruritis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eyelid ptosis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Foreign body sensation in eyes (Eye disorders) | 1 | 3 | 2 | 1 | 4 | 3 | 2
Iris adhesions (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Iris disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Iritis (Eye disorders) | 0 | 2 | 0 | 1 | 1 | 3 | 4
Keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 3 | 1 | 0 | 0 | 0 | 1
Macular degeneration (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Narrow anterior chamber angle (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ocular discomfort (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2
Ocular hyperaemia (Eye disorders) | 4 | 3 | 2 | 1 | 4 | 4 | 4
Optic disc haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 2 | 0 | 1 | 1 | 1 | 3
Photopsia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Posterior capsule opacification (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Punctate keratitis (Eye disorders) | 3 | 1 | 2 | 1 | 2 | 0 | 0
Recession of chamber angle of eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Trichiasis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Large intestinal polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Instillation site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 1 | 0
Upper respiratory track infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 1 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eosinophil count increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intraocular pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 3
Hypercholesterolemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Visual field defect (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bladder prolapse (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperemia (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-02-19): https://cdn.clinicaltrials.gov/large-docs/46/NCT02371746/Prot_000.pdf
  • Statistical Analysis Plan (2015-09-23): https://cdn.clinicaltrials.gov/large-docs/46/NCT02371746/SAP_001.pdf